CLINICAL TRIAL: NCT00331292
Title: A Study to Identify a Transcriptomic Profile Indicative of Cycle AMP Pathway Activation in the Lung
Brief Title: A Methodology Study To Look At Genes In Lung Cells And Tissue From Asthmatic Patients
Status: Terminated | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Other Study IDs: CRB100706
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Asthma
Keywords: Asthma bronchoscopy
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The primary goal of this study is to identify a gene or panel of genes which are differentially expressed in lung cells and tissue from asthmatic patients following administration of Ipratropium bromide and eiTher nebulised Albuterol or saline. Each subject in this study will undergo two bronchoscopies.

ELIGIBILITY:
Inclusion criteria:

* Have a history of intermittant asthma.
* Have asthma symptoms less than once per week.
* Have no other significant disease.
* Do not take regular oral or inhaled steroids.
* Are a non-smoker for the past 12 months with a pack history of less than 5 years.

Exclusion criteria:

* Have a history of drug or alcohol abuse.
* Have poorly controlled asthma or a history of life-threatening asthma.
* Have a history of hypersensitivity to bronchodilators.
* Are unable to abstain from inhaled steroids from 14 days prior to the first study visit until completion of the study.
* Have received oral steroids within 3 months of study entry.
* Have been hospitalized for your asthma within 3 months of study entry.
* Have had treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30
Dates: Start 2006-08

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Philadelphia, Pennsylvania, United States